CLINICAL TRIAL: NCT00734344
Title: Pilot Study of Raltegravir/Tenofovir/Emtricitabine Versus Efavirenz/Tenofovir/Emtricitabine for Adults With Acute HIV-1 Infection: Exploring the Role of Integrase Inhibition in Early HIV Pathogenesis
Brief Title: Pilot Study of Raltegravir/Truvada Versus Efavirenz/Truvada for Adults With Acute IV-1 Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Sonya Heath, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F080416007
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-04

CONDITIONS: Acute HIV Infection
MeSH Terms: interventions — Raltegravir Potassium; efavirenz

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): Raltegravir plus Truvada
  Interventions: Drug: Raltegravir; Drug: Emtricitibine; Drug: Tenofovir disoproxil twice daily
- Arm 2 (Active Comparator): Efavirenz plus Truvada
  Interventions: Drug: Efavirenz; Drug: Emtricitibine; Drug: Tenofovir disoproxil once daily

INTERVENTIONS:
Drug: Raltegravir — Raltegravir 400 mg. BID
  Arms: Arm 1
Drug: Efavirenz — 600 mg once daily
  Arms: Arm 2
Drug: Emtricitibine — 200mg once daily
Drug: Tenofovir disoproxil once daily — 300mg once daily
  Arms: Arm 2
Drug: Tenofovir disoproxil twice daily — 300mg twice daily
  Arms: Arm 1

SUMMARY:
This is a single-site, investigator-initiated, open-label, randomized/controlled clinical trial to compare the viral load response in plasma (and, in a subset of subjects, in gastrointestinal lymphoid tissue reservoirs) in subjects with acute/early HIV-1 infection treated with 12 weeks of raltegravir-based versus efavirenz-based ART (each combined with tenofovir/emtricitabine). Subjects will receive a self-limited course of therapy rather than a commitment to life-long HAART, as has been the experimental approach in a variety of clinical protocols in the United States and Europe. Subjects will complete a 12 week course of therapy, and those who meet treatment-response and safety criteria will then undergo a similarly intensive period of virology and immunology monitoring to compare the timing and dynamics of any observed virologic rebound following the treatment intervention.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 19 years of age or older who meet the NIH Acute Infection and Early Disease Research Program (AIEDRP) definition of acute or early HIV-1 infection. Briefly, acute HIV-1 infection is defined as > 5000 copies per milliliter of HIV RNA and one of the following documented within a 7 day period of the initial positive PCR-based assay: 1) a negative HIV-1 EIA or 2) a positive EIA with a negative or indeterminant HIV-1 Western Blot test (interpreted based on current CDC guidelines). For the purposes of this protocol, early HIV-1 infection is defined as detectable HIV RNA by PCR-based assay, a positive HIV EIA, a positive HIV-1 Western blot, and one of the following: 1) a documented negative HIV EIA in the preceding 6 months or 2) an HIV detuned EIA standardized optical density measurement (defined as sample OD - negative control OD/ positive control OD) of < 1.0 within 14 days of the positive HIV EIA (consistent with acute infection occurring in the past 120 days).

Exclusion Criteria:

* Lack consistent evidence of seroconversion or documented appropriate antibody testing for persistent HIV infection during the screening and early follow-up period.
* Prior receipt of antiretroviral therapy.
* Serum creatinine > 2.0 x upper limit of normal or a calculated creatinine clearance at time of screening < 30 mL/min (and 0.85X this value for females).
* Alkaline phosphatase >5 x upper limit of normal.
* AST (SGOT) and ALT (SGPT) > 5 x upper limit of normal. Repeat of a laboratory screening test will be allowed for test results that are unexpected based on documented prior laboratory results or to monitor declining trends that may relate to the primary retroviral syndrome.
* Have any severe medical illness that the investigators feel will interfere with the ability to take therapy or that will result in making therapy too risky for the subject. This includes active tuberculosis treatment, severe liver disease due to alcoholism or viral hepatitis, or unstable cardiovascular or cerebrovascular disease.
* Have significant psychiatric illness or ongoing substance abuse that, in the opinion of the investigators, would compromise the ability of the subject to provide adequate informed consent or to adhere to the study procedures safely and consistently.
* Women who are pregnant or actively breastfeeding at the time of screening.
* Men or women who are actively attempting to become pregnant, or who are unable or unwilling to institute adequate birth control measures during the entire course of this treatment protocol.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-09; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonya Heath, M. D., Principal Investigator — Department of Medicine Divison of Infectious Disease
Locations (1):
- UAB 1917 Clinic, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Raltegravir plus Truvada
  Raltegravir, tenofovir, emtricitibine: Raltegravir 400 mg. BID combined with tenofovir 300 mg and emtricitibine 200 mg once daily
- Arm 2: Efavirenz plus Truvada
  Efavirenz plus tenofovir with emtricitibine: efavirenz 600 mg once daily combined with tenofovir 300mg and emtricitibine 200mg once daily
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 9 | 7 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Mean White Blood Cell Count Between Treatment Groups at 2 Months
Description: Mean WBC count for all subjects as determined by standard lab procedures at 2 months after starting study drug as well as range. The normal number of WBCs in the blood is 4,500-10,000 white blood cells per microliter (mcL).
Time Frame: baseline to 2 months
Population: Raltegravir plus Truvada arm, there was no data for 1 subject because either the subject missed a visit or chose not to stop therapy.
Measure: Mean (Full Range); unit: white blood cells per microliter (mcL).
Groups:
- Raltegravir Plus Truvada: Raltegravir, Truvada (tenofovir, emtricitibine): Raltegravir 400 mg. BID combined with tenofovir 300 mg and emtricitibine 200 mg once daily
- Efavirenz Plus Truvada: Efavirenz plus Truvada (tenofovir, emtricitibine): tenofovir with emtricitibine: efavirenz 600 mg once daily combined with tenofovir 300mg and emtricitibine 200mg once daily
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 8 | 9
white blood cells per microliter (mcL). | 5904 [2450 to 139600] | 4918 [2870 to 6650]

2. Primary Outcome: Mean White Blood Cell Count Between Treatment Groups at 4 Months
Description: Mean WBC count of all subjects as determined by standard lab procedures at 4 months after starting study drug as well as range. The normal number of WBCs in the blood is 4,500-10,000 white blood cells per microliter (mcL).
Time Frame: 4 months post baseline
Population: In the Raltegravir plus Truvada arm, there was no data for 1 subject because either the subject missed a visit or chose not to stop therapy; in the Efavirenz plus Tuvada arm, there was no date for 3 subjects because either the subjects missed a visit or chose not to stop therapy
Measure: Mean (Full Range); unit: white blood cells per microliter (mcL).
Groups:
- Raltegravir Plus Truvada: Raltegravir, tenofovir, emtricitibine: Raltegravir 400 mg. BID combined with tenofovir 300 mg and emtricitibine 200 mg once daily
- Efavirenz Plus Truvada: Efavirenz plus tenofovir with emtricitibine: efavirenz 600 mg once daily combined with tenofovir 300mg and emtricitibine 200mg once daily
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 8 | 5
white blood cells per microliter (mcL). | 5850 [2840 to 12640] | 4948 [3230 to 6370]

3. Primary Outcome: Mean White Blood Cell Count Between Treatment Groups at 6 Months
Description: Mean WBC count of all subjects as determined by standard lab procedures at 6 months after starting study drug as well as range. The normal number of WBCs in the blood is 4,500-10,000 white blood cells per microliter (mcL).
Time Frame: 6 months after baseline
Population: In the Raltegravir plus Truvada arm, there was no data for 1 subject because either the subject missed a visit or chose not to stop therapy; in the Efavirenz plus Tuvada arm, there was no date for 4 subjects because either the subjects missed a visit or chose not to stop therapy
Measure: Mean (Full Range); unit: white blood cells per microliter (mcL).
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 8 | 5
white blood cells per microliter (mcL). | 5219 [2860 to 8630] | 4522 [3230 to 5530]

4. Primary Outcome: Mean White Blood Cell Count Between Treatment Groups at 8 Months
Description: Mean WBC count of all subjects as determined by standard lab procedures at 8 months after starting study drug as well as range. The normal number of WBCs in the blood is 4,500-10,000 white blood cells per microliter (mcL).
Time Frame: 8 months after baseline
Population: In the Raltegravir plus Truvada arm, there was no data for 3 subjects because either the subject missed a visit or chose not to stop therapy; in the Efavirenz plus Tuvada arm, there was no date for 4 subjects because either the subjects missed a visit or chose not to stop therapy
Measure: Mean (Full Range); unit: white blood cells per microliter (mcL).
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 6 | 5
white blood cells per microliter (mcL). | 6240 [3540 to 10800] | 4607 [2820 to 5820]

5. Primary Outcome: Mean White Blood Cell Count Between Treatment Groups at 10 Months
Description: Mean WBC count of all subjects as determined by standard lab procedures at 10 months after starting study drug as well as range. The normal number of WBCs in the blood is 4,500-10,000 white blood cells per microliter (mcL).
Time Frame: 10 months after baseline
Population: In the Raltegravir plus Truvada arm, there was no data for 7 subjects because either the subject missed a visit or chose not to stop therapy; in the Efavirenz plus Tuvada arm, there was no date for 7 subjects because either the subjects missed a visit or chose not to stop therapy
Measure: Mean (Full Range); unit: white blood cells per microliter (mcL).
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 2 | 2
white blood cells per microliter (mcL). | 5230 [5030 to 5430] | 4615 [4420 to 4810]

6. Primary Outcome: Mean White Blood Cell Count Between Treatment Groups at 12 Months
Description: Mean WBC count of all subjects as determined by standard lab procedures at 12 months after starting study drug as well as range. The normal number of WBCs in the blood is 4,500-10,000 white blood cells per microliter (mcL).
Time Frame: 12 months after baseline
Population: In the Raltegravir plus Truvada arm, there was no data for 6 subjects because either the subject missed a visit or chose not to stop therapy; in the Efavirenz plus Tuvada arm, there was no date for 5 subjects because either the subjects missed a visit or chose not to stop therapy
Measure: Mean (Full Range); unit: white blood cells per microliter (mcL).
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 3 | 4
white blood cells per microliter (mcL). | 6320 [4950 to 7470] | 4868 [3980 to 5710]

7. Primary Outcome: Mean White Blood Cell Count Between Treatment Groups at 14 Months
Description: Mean WBC count of all subjects as determined by standard lab procedures at 14 months after starting study drug as well as range. The normal number of WBCs in the blood is 4,500-10,000 white blood cells per microliter (mcL).
Time Frame: 14 months after baseline
Population: In the Raltegravir plus Truvada arm, there was no data for 8 subjects because either the subject missed a visit or chose not to stop therapy; in the Efavirenz plus Tuvada arm, there was no date for 6 subjects because either the subjects missed a visit or chose not to stop therapy
Measure: Mean (Full Range); unit: white blood cells per microliter (mcL).
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 1 | 3
white blood cells per microliter (mcL). | 3180 [3180 to 3180] | 4903 [4360 to 5840]

8. Primary Outcome: Mean Hematocrit Between Treatment Groups at 2 Months
Description: Mean hematocrit of all subjects at 2 months after starting study drug. The hematocrit, also known as packed cell volume (PCV) or erythrocyte volume fraction (EVF), is the volume percentage (%) of red blood cells in blood. It is normally 45% for men and 40% for women.
Time Frame: 2 months after baseline
Population: In the Raltegravir plus Truvada arm, there was no data for 1 subject because either the subject missed a visit or chose not to stop therapy
Measure: Mean (Full Range); unit: percentage
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 8 | 9
percentage | 41.5 [36 to 46] | 41.8 [37 to 50]

9. Primary Outcome: Mean Hematocrit Between Treatment Groups at 4 Months
Description: Mean hematocrit of all subjects at 4 months after starting study drug. The hematocrit, also known as packed cell volume (PCV) or erythrocyte volume fraction (EVF), is the volume percentage (%) of red blood cells in blood. It is normally 45% for men and 40% for women.
Time Frame: 4 months after baseline
Population: as for outcome 3
Measure: Mean (Full Range); unit: percentage
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 8 | 5
percentage | 41.4 [34 to 48] | 43 [37 to 51]

10. Primary Outcome: Mean Hematocrit Between Treatment Groups at 6 Months
Description: Mean hematocrit of all subjects at 6 months after starting study drug. The hematocrit, also known as packed cell volume (PCV) or erythrocyte volume fraction (EVF), is the volume percentage (%) of red blood cells in blood. It is normally 45% for men and 40% for women.
Time Frame: 6 months after baseline
Population: as for outcome 3
Measure: Mean (Full Range); unit: percentage
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 8 | 5
percentage | 42.1 [36 to 47] | 39.8 [35 to 50]

11. Primary Outcome: Mean Hematocrit Between Treatment Groups at 8 Months
Description: Mean hematocrit of all subjects at 8 months after starting study drug. The hematocrit, also known as packed cell volume (PCV) or erythrocyte volume fraction (EVF), is the volume percentage (%) of red blood cells in blood. It is normally 45% for men and 40% for women.
Time Frame: 8 months after baseline
Population: In the Raltegravir plus Truvada arm, there was no data for 3 subjects because either the subject missed a visit or chose not to stop therapy; in the Efavirenz plus Tuvada arm, there was no date for 3 subjects because either the subjects missed a visit or chose not to stop therapy
Measure: Mean (Full Range); unit: percentage
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 6 | 6
percentage | 40.3 [37 to 45] | 41.2 [36 to 51]

12. Primary Outcome: Mean Hematocrit Between Treatment Groups at 10 Months
Description: Mean hematocrit of all subjects at 10 months after starting study drug. The hematocrit, also known as packed cell volume (PCV) or erythrocyte volume fraction (EVF), is the volume percentage (%) of red blood cells in blood. It is normally 45% for men and 40% for women.
Time Frame: 10 months after baseline
Population: as for outcome 5
Measure: Mean (Full Range); unit: percentage
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 2 | 2
percentage | 45 [42 to 48] | 38 [37 to 39]

13. Primary Outcome: Mean Hematocrit Between Treatment Groups at 12 Months
Description: Mean hematocrit of all subjects at 12 months after starting study drug. The hematocrit, also known as packed cell volume (PCV) or erythrocyte volume fraction (EVF), is the volume percentage (%) of red blood cells in blood. It is normally 45% for men and 40% for women.
Time Frame: 12 months after baseline
Population: as for outcome 6
Measure: Mean (Full Range); unit: percentage
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 3 | 4
percentage | 41 [37 to 45] | 43.5 [39 to 52]

14. Primary Outcome: Mean Hematocrit Between Treatment Groups at 14 Months
Description: Mean hematocrit of all subjects at 14 months after starting study drug. The hematocrit, also known as packed cell volume (PCV) or erythrocyte volume fraction (EVF), is the volume percentage (%) of red blood cells in blood. It is normally 45% for men and 40% for women.
Time Frame: 14 months after baseline
Population: as for outcome 7
Measure: Mean (Full Range); unit: percentage
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 1 | 3
percentage | 36 [36 to 36] | 39.7 [39 to 40]

15. Primary Outcome: Mean Platelet Count Between Treatment Groups at 2 Months
Description: The mean platelet count between treament groups at 2 months after starting study drug. The calculated number of platelets in a volume of blood, usually expressed as platelets per cubic millimeter (cmm) of whole blood. Platelets are the smallest cell-like structures in the blood and are important for blood clotting and plugging damaged blood vessels. Platelet counts are usually done by laboratory machines that also count other blood elements such as the white and red cells. They can also be counted by use of a microscope. Normal platelet counts are in the range of 150,000 to 400,000 per microliter (or 150 - 400 x 100 per liter).
Time Frame: 2 months after baseline
Population: In the Raltegravir plus Truvada arm, there was no data for 1 subject because either the subject missed a visit or chose not to stop therapy; in the Efavirenz plus Tuvada arm
Measure: Mean (Full Range); unit: count per microliter
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 8 | 9
count per microliter | 232600 [166200 to 336100] | 225600 [154700 to 306800]

16. Primary Outcome: Mean Platelet Count Between Treatment Groups at 4 Months
Description: The mean platelet count between treatment groups at 4 months after starting study drug. The calculated number of platelets in a volume of blood, usually expressed as platelets per cubic millimeter (cmm) of whole blood. Platelets are the smallest cell-like structures in the blood and are important for blood clotting and plugging damaged blood vessels. Platelet counts are usually done by laboratory machines that also count other blood elements such as the white and red cells. They can also be counted by use of a microscope. Normal platelet counts are in the range of 150,000 to 400,000 per microliter (or 150 - 400 x 109 per liter).
Time Frame: 4 months after baseline
Population: as for outcome 3
Measure: Mean (Full Range); unit: count per microliter
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 8 | 5
count per microliter | 210800 [157600 to 343200] | 197300 [144600 to 263900]

17. Primary Outcome: Mean Platelet Count Between Treatment Groups at 6 Months
Description: The mean platelet count between treatment groups at 6 months after starting study drug. The calculated number of platelets in a volume of blood, usually expressed as platelets per cubic millimeter (cmm) of whole blood. Platelets are the smallest cell-like structures in the blood and are important for blood clotting and plugging damaged blood vessels. Platelet counts are usually done by laboratory machines that also count other blood elements such as the white and red cells. They can also be counted by use of a microscope. Normal platelet counts are in the range of 150,000 to 400,000 per microliter (or 150 - 400 x 109 per liter).
Time Frame: 6 months after baseline
Population: as for outcome 3
Measure: Mean (Full Range); unit: count per microliter
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 8 | 5
count per microliter | 230000 [162600 to 307000] | 224800 [129700 to 309100]

18. Primary Outcome: Mean Platelet Count Between Treatment Groups at 8 Months
Description: The mean platelet count between treatment groups at 8 months after starting study drug. The calculated number of platelets in a volume of blood, usually expressed as platelets per cubic millimeter (cmm) of whole blood. Platelets are the smallest cell-like structures in the blood and are important for blood clotting and plugging damaged blood vessels. Platelet counts are usually done by laboratory machines that also count other blood elements such as the white and red cells. They can also be counted by use of a microscope. Normal platelet counts are in the range of 150,000 to 400,000 per microliter (or 150 - 400 x 109 per liter).
Time Frame: 8 months after baseline
Population: as for outcome 11
Measure: Mean (Full Range); unit: count per microliter
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 6 | 6
count per microliter | 215700 [108000 to 333200] | 208100 [131200 to 265900]

19. Primary Outcome: Mean Platelet Count Between Treatment Groups at 10 Months
Description: The mean platelet count between treatment groups at 10 months after starting study drug. The calculated number of platelets in a volume of blood, usually expressed as platelets per cubic millimeter (cmm) of whole blood. Platelets are the smallest cell-like structures in the blood and are important for blood clotting and plugging damaged blood vessels. Platelet counts are usually done by laboratory machines that also count other blood elements such as the white and red cells. They can also be counted by use of a microscope. Normal platelet counts are in the range of 150,000 to 400,000 per microliter (or 150 - 400 x 109 per liter).
Time Frame: 10 months after baseline
Population: as for outcome 5
Measure: Mean (Full Range); unit: count per microliter
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 2 | 2
count per microliter | 193500 [187600 to 199500] | 243300 [196600 to 290100]

20. Primary Outcome: Mean Platelet Count Between Treatment Groups at 12 Months
Description: The mean platelet count between treatment groups at 12 months after starting study drug. The calculated number of platelets in a volume of blood, usually expressed as platelets per cubic millimeter (cmm) of whole blood. Platelets are the smallest cell-like structures in the blood and are important for blood clotting and plugging damaged blood vessels. Platelet counts are usually done by laboratory machines that also count other blood elements such as the white and red cells. They can also be counted by use of a microscope. Normal platelet counts are in the range of 150,000 to 400,000 per microliter (or 150 - 400 x 109 per liter).
Time Frame: 12 months after baseline
Population: as for outcome 6
Measure: Mean (Full Range); unit: count per microliter
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 3 | 4
count per microliter | 255600 [207700 to 318600] | 185500 [144600 to 216900]

21. Primary Outcome: Mean Platelet Count Between Treatment Groups at 14 Months
Description: The mean platelet count between treatment groups at 14 months after starting study drug. The calculated number of platelets in a volume of blood, usually expressed as platelets per cubic millimeter (cmm) of whole blood. Platelets are the smallest cell-like structures in the blood and are important for blood clotting and plugging damaged blood vessels. Platelet counts are usually done by laboratory machines that also count other blood elements such as the white and red cells. They can also be counted by use of a microscope. Normal platelet counts are in the range of 150,000 to 400,000 per microliter (or 150 - 400 x 109 per liter).
Time Frame: 4 months after baseline
Population: as for outcome 7
Measure: Mean (Full Range); unit: count per microliter
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 1 | 3
count per microliter | 217400 [217400 to 217400] | 216800 [191400 to 247000]

22. Primary Outcome: Mean CD4 Count Between Treatment Groups at 1 Months
Description: Mean CD4 count between groups 1 month after starting study drug. CD4 cells are types of white blood cells called T lymphocytes or T cells that fight infection. CD4 counts are most often used to evaluate the immune system of a person diagnosed with a human immunodeficiency virus (HIV) infection to help stage and monitor progression of the disease and monitor effectiveness of antiretroviral treatment. A CD4 count is typically reported as an absolute level or count of cells (expressed as cells per cubic millimeter of blood). A normal CD4 count ranges from 410-1,590 cells/mm3. Sometimes results are expressed as a percent of total lymphocytes (CD4 percent).
Time Frame: 1 month after baseline
Measure: Mean (Full Range); unit: cells/mm3
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 9 | 9
cells/mm3 | 629.1 [345 to 1157] | 535 [370 to 773]

23. Primary Outcome: Mean CD4 Count Between Treatment Groups at 2 Months
Description: Mean CD4 count between groups 2 months after starting study drug. CD4 cells are types of white blood cells called T lymphocytes or T cells that fight infection. CD4 counts are most often used to evaluate the immune system of a person diagnosed with a human immunodeficiency virus (HIV) infection to help stage and monitor progression of the disease and monitor effectiveness of antiretroviral treatment. A CD4 count is typically reported as an absolute level or count of cells (expressed as cells per cubic millimeter of blood). A normal CD4 count ranges from 410-1,590 cells/mm3 in adults and teens. Sometimes results are expressed as a percent of total lymphocytes (CD4 percent).
Time Frame: 2 months after baseline
Population: In the Raltegravir plus Truvada arm, there was no data for 1 subject because either the subject missed a visit or chose not to stop therapy; in the Efavirenz plus Tuvada arm, there was no date for 1 subject because either the subjects missed a visit or chose not to stop therapy
Measure: Mean (Full Range); unit: cells/mm3
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 8 | 8
cells/mm3 | 703.1 [300 to 1541] | 527.2 [336 to 787]

24. Primary Outcome: Mean CD4 Count Between Treatment Groups at 3 Months
Description: Mean CD4 count between groups 3 months after starting study drug. CD4 cells are types of white blood cells called T lymphocytes or T cells that fight infection. CD4 counts are most often used to evaluate the immune system of a person diagnosed with a human immunodeficiency virus (HIV) infection to help stage and monitor progression of the disease and monitor effectiveness of antiretroviral treatment. A CD4 count is typically reported as an absolute level or count of cells (expressed as cells per cubic millimeter of blood). A normal CD4 count ranges from 410-1,590 cells/mm3 in adults and teens. Sometimes results are expressed as a percent of total lymphocytes (CD4 percent).
Time Frame: 3 months after baseline
Population: as for outcome 2
Measure: Mean (Full Range); unit: cells/mm3
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 8 | 6
cells/mm3 | 716.4 [399 to 1251] | 671.7 [485 to 903]

25. Primary Outcome: Mean CD4 Count Between Treatment Groups at 4 Months
Description: Mean CD4 count between groups 4 months after starting study drug. CD4 cells are types of white blood cells called T lymphocytes or T cells that fight infection. CD4 counts are most often used to evaluate the immune system of a person diagnosed with a human immunodeficiency virus (HIV) infection to help stage and monitor progression of the disease and monitor effectiveness of antiretroviral treatment. A CD4 count is typically reported as an absolute level or count of cells (expressed as cells per cubic millimeter of blood). A normal CD4 count ranges from 410-1,590 cells/mm3 in adults and teens. Sometimes results are expressed as a percent of total lymphocytes (CD4 percent).
Time Frame: 4 months after baseline
Population: In the Raltegravir plus Truvada arm, there was no data for 4 subjects because either the subject missed a visit or chose not to stop therapy; in the Efavirenz plus Tuvada arm, there was no date for 7 subjects because either the subjects missed a visit or chose not to stop therapy
Measure: Mean (Full Range); unit: cells/mm3
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 5 | 2
cells/mm3 | 617.2 [362 to 901] | 646.5 [589 to 704]

26. Primary Outcome: Mean CD4 Count Between Treatment Groups at 5 Months
Description: Mean CD4 count between groups 5 months after starting study drug. CD4 cells are types of white blood cells called T lymphocytes or T cells that fight infection. CD4 counts are most often used to evaluate the immune system of a person diagnosed with a human immunodeficiency virus (HIV) infection to help stage and monitor progression of the disease and monitor effectiveness of antiretroviral treatment. A CD4 count is typically reported as an absolute level or count of cells (expressed as cells per cubic millimeter of blood). A normal CD4 count ranges from 410-1,590 cells/mm3 in adults and teens. Sometimes results are expressed as a percent of total lymphocytes (CD4 percent).
Time Frame: 5 months after baseline
Population: as for outcome 4
Measure: Mean (Full Range); unit: cells/mm3
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 6 | 5
cells/mm3 | 805.7 [446 to 1991] | 539.6 [386 to 711]

27. Primary Outcome: Mean CD4 Count Between Treatment Groups at 6 Months
Description: Mean CD4 count between groups 6 months after starting study drug. CD4 cells are types of white blood cells called T lymphocytes or T cells that fight infection. CD4 counts are most often used to evaluate the immune system of a person diagnosed with a human immunodeficiency virus (HIV) infection to help stage and monitor progression of the disease and monitor effectiveness of antiretroviral treatment. A CD4 count is typically reported as an absolute level or count of cells (expressed as cells per cubic millimeter of blood). A normal CD4 count ranges from 410-1,590 cells/mm3 in adults and teens. Sometimes results are expressed as a percent of total lymphocytes (CD4 percent).
Time Frame: 6 months after baseline
Population: as for outcome 25
Measure: Mean (Full Range); unit: cells/mm3
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 5 | 2
cells/mm3 | 652.2 [435 to 986] | 673.5 [665 to 682]

28. Primary Outcome: Mean CD4 Count Between Treatment Groups at 7 Months
Description: Mean CD4 count between groups 7 months after starting study drug. CD4 cells are types of white blood cells called T lymphocytes or T cells that fight infection. CD4 counts are most often used to evaluate the immune system of a person diagnosed with a human immunodeficiency virus (HIV) infection to help stage and monitor progression of the disease and monitor effectiveness of antiretroviral treatment. A CD4 count is typically reported as an absolute level or count of cells (expressed as cells per cubic millimeter of blood). A normal CD4 count ranges from 410-1,590 cells/mm3 in adults and teens. Sometimes results are expressed as a percent of total lymphocytes (CD4 percent).
Time Frame: 7 months after baseline
Population: In the Raltegravir plus Truvada arm, there was no data for 5 subjects because either the subject missed a visit or chose not to stop therapy; in the Efavirenz plus Tuvada arm, there was no date for 7 subjects because either the subjects missed a visit or chose not to stop therapy
Measure: Mean (Full Range); unit: cells/mm3
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 4 | 2
cells/mm3 | 504 [300 to 662] | 552.5 [467 to 638]

29. Primary Outcome: Mean CD4 Count Between Treatment Groups at 8 Months
Description: Mean CD4 count between groups 8 months after starting study drug. CD4 cells are types of white blood cells called T lymphocytes or T cells that fight infection. CD4 counts are most often used to evaluate the immune system of a person diagnosed with a human immunodeficiency virus (HIV) infection to help stage and monitor progression of the disease and monitor effectiveness of antiretroviral treatment. A CD4 count is typically reported as an absolute level or count of cells (expressed as cells per cubic millimeter of blood). A normal CD4 count ranges from 410-1,590 cells/mm3 in adults and teens. Sometimes results are expressed as a percent of total lymphocytes (CD4 percent).
Time Frame: 8 months after baseline
Population: as for outcome 28
Measure: Mean (Full Range); unit: cells/mm3
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 4 | 2
cells/mm3 | 464.5 [365 to 628] | 586.5 [485 to 688]

30. Primary Outcome: Mean CD4 Count Between Treatment Groups at 9 Months
Description: Mean CD4 count between groups 9 months after starting study drug. CD4 cells are types of white blood cells called T lymphocytes or T cells that fight infection. CD4 counts are most often used to evaluate the immune system of a person diagnosed with a human immunodeficiency virus (HIV) infection to help stage and monitor progression of the disease and monitor effectiveness of antiretroviral treatment. A CD4 count is typically reported as an absolute level or count of cells (expressed as cells per cubic millimeter of blood). A normal CD4 count ranges from 410-1,590 cells/mm3 in adults and teens. Sometimes results are expressed as a percent of total lymphocytes (CD4 percent).
Time Frame: 9 months after baseline
Population: In the Raltegravir plus Truvada arm, there was no data for 8 subjects because either the subject missed a visit or chose not to stop therapy; in the Efavirenz plus Tuvada arm, there was no date for 8 subjects because either the subjects missed a visit or chose not to stop therapy
Measure: Mean (Full Range); unit: cells/mm3
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 1 | 1
cells/mm3 | 306 [306 to 306] | 571 [571 to 571]

31. Primary Outcome: Mean CD4 Count Between Treatment Groups at 10 Months
Description: Mean CD4 count between groups 10 months after starting study drug. CD4 cells are types of white blood cells called T lymphocytes or T cells that fight infection. CD4 counts are most often used to evaluate the immune system of a person diagnosed with a human immunodeficiency virus (HIV) infection to help stage and monitor progression of the disease and monitor effectiveness of antiretroviral treatment. A CD4 count is typically reported as an absolute level or count of cells (expressed as cells per cubic millimeter of blood). A normal CD4 count ranges from 410-1,590 cells/mm3 in adults and teens. Sometimes results are expressed as a percent of total lymphocytes (CD4 percent).
Time Frame: 10 months after baseline
Population: In the Raltegravir plus Truvada arm, there was no data for 8 subjects because either the subject missed a visit or chose not to stop therapy; in the Efavirenz plus Tuvada arm, there was no date for 7 subjects because either the subjects missed a visit or chose not to stop therapy
Measure: Mean (Full Range); unit: cells/mm3
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 1 | 2
cells/mm3 | 469 [469 to 469] | 571.5 [561 to 582]

32. Primary Outcome: Mean CD4 Count Between Treatment Groups at 11 Months
Description: Mean CD4 count between groups 11 months after of starting study drug. CD4 cells are types of white blood cells called T lymphocytes or T cells that fight infection. CD4 counts are most often used to evaluate the immune system of a person diagnosed with a human immunodeficiency virus (HIV) infection to help stage and monitor progression of the disease and monitor effectiveness of antiretroviral treatment. A CD4 count is typically reported as an absolute level or count of cells (expressed as cells per cubic millimeter of blood). A normal CD4 count ranges from 410-1,590 cells/mm3 in adults and teens. Sometimes results are expressed as a percent of total lymphocytes (CD4 percent).
Time Frame: 11 months after baseline
Population: In the Raltegravir plus Truvada arm, there was no data for 9 subjects because either the subject missed a visit or chose not to stop therapy; in the Efavirenz plus Tuvada arm, there was no date for 9 subjects because either the subjects missed a visit or chose not to stop therapy
Measure: Mean (Full Range); unit: cells/mm3
Arm/Group | Raltegravir Plus Truvada | Efavirenz Plus Truvada
Number analyzed (Participants) | 1 | 0
cells/mm3 | 495 [495 to 495] |

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes